CLINICAL TRIAL: NCT07009938
Title: Long-Term Efficacy and Safety of Drug-Coated Balloon Angioplasty in Patients With Coronary Artery Disease and Type 2 Diabetes: A Multicenter, Prospective, Randomized Controlled Trial
Brief Title: DCB for CAD With Type 2 Diabetes
Acronym: DCBinT2DM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Chief Physician, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DCBinT2DM
Record Dates: First submitted 2025-05-25; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease; Diabete Type 2
Keywords: coronary artery disease; type 2 diabetes mellitus; drug-coated balloon; target lesion revascularization; major adverse cardiac events
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Drug-Eluting Stents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous coronary intervention using Drug-Coated Balloon (DCB) (Experimental): Percutaneous coronary intervention using Drug-Coated Balloon (DCB)
  Interventions: Device: Drug-Coated Balloon (DCB)
- Either Drug-Eluting Stent (DES) implantation group (Active Comparator): Percutaneous coronary intervention using Drug-Eluting Stent (DES) implantation
  Interventions: Device: Drug-Eluting Stent (DES) implantation

INTERVENTIONS:
Device: Drug-Coated Balloon (DCB) — Following lesion preparation (usually with a standard balloon), a drug-coated balloon is advanced to the target lesion. The balloon is inflated and maintained to allow effective drug transfer to the vessel wall.
  Arms: Percutaneous coronary intervention using Drug-Coated Balloon (DCB)
Device: Drug-Eluting Stent (DES) implantation — After coronary angiography identifies the target lesion, a DES is selected based on the vessel size. Post-deployment angiography is performed to confirm the result and check for complications.
  Arms: Either Drug-Eluting Stent (DES) implantation group

SUMMARY:
Patients with coronary artery disease (CAD) and type 2 diabetes mellitus (T2DM) often present with diffuse, complex lesions and a higher risk of in-stent restenosis after PCI. While drug-eluting stents (DES) remain the standard treatment, their long-term efficacy in diabetic patients is suboptimal. Drug-coated balloons (DCBs) offer a "leave nothing behind" strategy by delivering anti-proliferative drugs without permanent implants, potentially reducing restenosis and adverse events. Although DCBs have shown promise in selected lesion types, evidence in T2DM patients is limited, particularly from prospective, randomized trials. This study aims to evaluate the efficacy and safety of DCB angioplasty compared to conventional strategies in patients with CAD and T2DM, focusing on angiographic outcomes, symptom relief, and major adverse cardiovascular events.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) and type 2 diabetes mellitus (T2DM) often coexist, and the long-term hyperglycemic state and metabolic disorders in diabetic patients contribute to endothelial dysfunction and accelerated atherosclerosis. As a result, coronary lesions in T2DM patients tend to be more diffuse and complex, posing greater challenges to percutaneous coronary intervention (PCI). Although drug-eluting stents (DES) have significantly improved clinical outcomes, diabetic patients remain at higher risk for in-stent restenosis (ISR) and target lesion revascularization (TLR), negatively impacting long-term prognosis.

Drug-coated balloons (DCBs), a novel PCI technique, allow for rapid and effective delivery of anti-proliferative agents (e.g. paclitaxel or sirolimus) to the vessel wall without leaving behind a permanent implant. This "leave nothing behind" approach reduces the risk of chronic inflammation and stent-related complications. DCBs have shown promising results in non-diabetic populations, particularly in small vessel disease and bifurcation lesions. However, evidence supporting their use in T2DM patients remains limited, especially from prospective, randomized controlled trials. As such, whether DCBs can serve as a viable alternative to DES in this high-risk group remains an open question.

This study aims to evaluate the efficacy and safety of DCB angioplasty in patients with CAD and T2DM through a prospective, randomized controlled design. The study will focus on restenosis rates, improvement in angina symptoms, incidence of major adverse cardiovascular events (MACE), and patient-reported quality of life outcomes, providing a more individualized and evidence-based treatment approach for this challenging patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosed CAD with ≥70% stenosis in ≥1 coronary artery confirmed by coronary angiography
* Diagnosed type 2 diabetes (per WHO criteria)
* Target lesion suitable for DCB (diameter 2.0-4.0 mm, length ≤40 mm)
* Informed consent provided

Exclusion Criteria:

* Prior coronary artery bypass surgery or PCI with complications
* STEMI within 24 hours
* Severe hepatic/renal dysfunction
* Active bleeding or uncontrolled anticoagulation
* Allergy to DCB components
* Pregnancy or lactation
* Psychiatric conditions limiting compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Diameter Stenosis Rate | At 12 months after intervention
  Target Lesion Diameter Stenosis Rate refers to the percentage of narrowing at the target coronary lesion, calculated by comparing the minimal lumen diameter (MLD) at the lesion site with the reference vessel diameter (RVD), which was measured based on coronary angiography.

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | At 12 months after intervention
  A composite of cardiac death, myocardial infarction, target vessel revascularization, or stent thrombosis)
Angina Symptom Improvement | At baseline, 1, 3, 6 and 12 months after intervention
  Measured by Seattle Angina Questionnaire (SAQ) at baseline, 1, 3, and 6 months.
Changes in glycemic indices including glycated hemoglobin (HbA1c) | At 3, 6 and 12 months after intervention
  Changes in glycemic indices including glycated hemoglobin (HbA1c)
Glycemic indices | At 3, 6 and 12 months after intervention
  Changes in fasting blood glucose, and 2-hour postprandial blood glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Yidong Wei, PhD, Principal Investigator — Shanghai 10th People's Hospital
Locations (6):
- China (6):
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - Luoyang Central Hospital Affiliated to Zhengzhou University, Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou Uninversity, Zhengzhou, Henan
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - The Second People's Hospital of Yibin, Yibin, Sichuan
  - Ninghai First Hospital, Ningbo, Zhejiang